CLINICAL TRIAL: NCT00570128
Title: A 10-Week, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Donepezil Hydrochloride (Aricept®) in the Treatment of the Cognitive Dysfunction Exhibited by Children With Down Syndrome
Brief Title: Evaluating The Efficacy And Safety Of Donepezil Hydrochloride (HCl) (Aricept) In Treating Cognitive Dysfunction Exhibited By Children With Down Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-A001-219; A2501059 (Other: Pfizer)
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; trisomy 21
MeSH Terms: conditions — Down Syndrome | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donepezil HCl (Active Comparator)
  Interventions: Drug: Donepezil HCl
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil HCl — Blinded donepezil 2.5 milligram per day (mg/day) (2.5 milliliter per day [mL/day]) orally for participants with body weight (BW) 20 and less than (<) 25 kilogram (kg), 5 mg/day (5 mL/day) orally for participants with BW 25 to <50 kg, and 10 mg/day (10 mL/day) orally for participants with BW greater than or equal to (>=) 50 kg liquid formulation (1 milligram per 1 milliliter [1 mg/1 mL]) (titrated to 0.1 to 0.2 milligram per kilogram per day [mg/kg/day] based on BW).
  Other Names: Aricept
  Arms: Donepezil HCl
Drug: Placebo — Liquid formulation matched to active treatment for oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether donepezil HCl is effective and safe in improving cognitive dysfunction exhibited by children and adolescents with Down syndrome (DS). Effectiveness will be measured by rating communication, daily living skills, and social skills and relationships in subjects aged 10 to 17.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10 to 17 years old, weight more than or equal to 20 kg
* Male and female
* Vineland-II Adaptive Behavior Scales (VABS-II)/Parent/Caregiver Rating Form (PCRF) standard composite score greater than (>) 55
* Diagnosis of DS (trisomy 21) documented by chromosomal analysis (karyotyping). If such documentation is not available at screening, karyotyping will be performed with the screening labs and must be documented prior to baseline visit.
* Naïve to approved or unapproved cholinesterase inhibitors is preferred however, prior use of these medications is allowed, provided that the medication was discontinued at least 3 months prior to screening and that it was not discontinued for lack of tolerability or efficacy or for the sole purpose of enrolling the subject in the study.
* Subjects residing in the community
* Must be expected to complete all procedures scheduled during the Screening and Baseline visits including all efficacy and safety parameters.
* Must speak English and be verbal and able to be understood most of the time and must not use other forms of communication, signs, symbol boards or devices to supplement his/her communication ability
* Must have a parent or other reliable caregiver who agrees to accompany the subject to all clinic visits, provide information about the subject as required by the protocol, and ensure compliance with the medication schedule
* a Parent or Caregiver must be a constant and reliable informant with sufficient contact with the subject to have detailed knowledge of the subject's adaptive behavior in order to be able to complete the VABS-II/PCRF accurately. The same individual should complete the form at every visit.
* Should be in good general health with no medical conditions that are considered both clinically significant and unstable
* Clinical laboratory values within normal limits or abnormalities considered not clinically significant by the investigator and sponsor
* Stable Type I (insulin-dependent) or Type II diabetes are eligible provided they are monitored regularly prior to and during the study to ensure adequate glucose control (fasting blood glucose <140 milligram per deciliter (mg/dl) and glycosylated hemoglobin [hemoglobin A1c] <8 percent (%) at screening).
* Thyroid disease also may be included in the study provided they are euthyroid and stable on treatment for at least 3 months prior to screening.
* History of seizure disorder is allowed provided that subjects are on stable treatment for at least 3 months and have not had a seizure within the past 6 months.
* Independent in ambulation or ambulatory aided (example, walker or cane, wheelchair), vision and hearing (eyeglasses and/or hearing aid permissible) sufficient for achieving VABS-II/PCRF composite standard scores >55 and for cooperating with examinations and the Test of Verbal Expression and Reasoning (TOVER).

Exclusion Criteria:

* Ages <10 or >17 years
* Active or clinically significant conditions affecting absorption, distribution or metabolism of the study medication (example, inflammatory bowel disease, gastric or duodenal ulcers or severe lactose intolerance)
* Known hypersensitivity to piperidine derivatives or cholinesterase inhibitors
* Currently receiving cholinesterase inhibitors or who have received them in the 3 months prior to screening or with prior use >3 months prior to screening who stopped for lack of efficacy or tolerability
* No reliable parent or caregiver, or participants, or caregivers who are unwilling or unable to complete any of the outcome measures and fulfill the requirements of this study
* Clinically significant obstructive pulmonary disease or asthma untreated or not controlled by treatment within 3 months prior to screening
* Recent (less than or equal to 2 years) hematologic/oncologic disorders (mild anemia allowed)
* Evidence of active, clinically significant, and unstable gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease
* Current Diagnostic and Statistical Manual IV Text Revision (DSM-IV-TR) diagnosis of Major Depressive Disorder (MDD) or any current primary psychiatric diagnosis other than DS (as per DSM-IV)
* Any condition which would make the subject or the caregiver, in the opinion of the investigator, unsuitable for the study
* Unsuitability which includes female subjects who have begun menstruation and are thus of child-bearing potential, who may be sexually active and who are not practicing an effective means of birth control.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2007-11-16 (Actual); Primary Completion 2008-09-05 (Actual); Study Completion 2008-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Clinical Study Centers, L.L.C., Little Rock, Arkansas
  - Neufeld Medical Group, Inc., Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - University of California, Irvine Medical Center, Department of Pediatrics, Orange, California
  - UCSD Pediatric Pharmacology Research Unit, San Diego, California
  - Rocky Mountain Pediatrics, Lakewood, Colorado
  - Neuropsychiatric Research Center of South West Florida, Fort Myers, Florida
  - Miami Children's Hospital, Clinical Research Center, Miami, Florida
  - Community Research Foundation, Miami, Florida
  - Miami Children's Hospital, Brain Institute, Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - Lazlo J. Mate, MD, West Palm Beach, Florida
  - Child Neurology Associates, PC, Atlanta, Georgia
  - Medical Genetics and Neuro Development Center, Zionsville, Indiana
  - Hurley Medical Center, Flint, Michigan
  - Saint Mayr's Health Care, Grand Rapids, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Washington University School of Medicine, Division of Genetics and Genomic Medicine, St Louis, Missouri
  - Midwest Children's Health Research Institute, LLC, Lincoln, Nebraska
  - Clinical Research Center of New Jersey, Voorhees Township, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Metrohealth Medical Center, Division of Psychiatry, Cleveland, Ohio
  - Valko and Associates, Toledo, Ohio
  - Tulsa Clinical Research LLC, Tulsa, Oklahoma
  - Medical University of South Carolina, Division of Genetics and Developmental and Behavioral Pediatrics, Charleston, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Down Syndrome Clinic of Houston, Houston, Texas
  - Alamo City Clinical Research, LLC, San Antonio, Texas
  - Road Runner Research, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 35 centers in the United States during the period of 16 November 2007 to 05 September 2008.
Groups:
- Donepezil HCl: Blinded donepezil hydrochloride (HCl) 2.5 milligram per day (mg/day) (2.5 milliliter per day [mL/day]) orally for participants with body weight (BW) 20 and less than (<) 25 kilogram (kg), 5 mg/day (5 mL/day) orally for participants with BW 25 to <50 kg, and 10 mg/day (10 mL/day) orally for participants with BW greater than or equal to (>=) 50 kg liquid formulation (1 milligram per 1 milliliter [1 mg/1 mL]) (titrated to 0.1 to 0.2 milligram per kilogram per day [mg/kg/day] based on BW).
Period: Overall Study
Arm/Group | Donepezil HCl | Placebo
Started | 64 | 65
Intent to Treat (ITT) Population | 62 | 65
Completed | 60 | 65
Not Completed | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Donepezil HCl: Blinded donepezil HCl 2.5 mg/day (2.5 mL/day) orally for participants with BW 20 and <25 kg, 5 mg/day (5 mL/day) orally for participants with BW 25 to <50 kg, and 10 mg/day (10 mL/day) orally for participants with BW >=50 kg liquid formulation (1 mg/1 mL) (titrated to 0.1 to 0.2 mg/kg/day based on BW).
- Total: Total of all reporting groups
Arm/Group | Donepezil HCl | Placebo | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.0 (2.3) | 13.0 (2.1) | 13.0 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 35 | 63
  Male | 36 | 30 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 54 | 57 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in V-Scale Composite Score (Sum of 9 Sub-Domains) of Vineland Adaptive Behavior Scales Second Edition-Parent Caregiver Rating Form (VABS-II/PCRF) at Week 10-Last Observation Carried Forward (LOCF)
Description: The VABS-II/PCRF instrument was used in this study to assess 3 domains (each with 3 sub-domains): communication (sub-domains: receptive, expressive, and writing), daily living skills (sub-domains: personal, domestic, community), and socialization (sub-domains: interpersonal relationships, play/leisure time, coping skills). Raw scores (2=always present, 1=sometimes present, 0=seldom or never present) rated by the parent/caregiver from each sub-domain were converted to standardized scores called V-scores, which are based on age and a national sample of normal children. Each sub-domain v-scale score ranged from 1 (weakness) to 24 (strength). V-scores for the 9 sub-domains were summed to obtain a composite V-score ranging from 9 to 216. Higher scores indicate a higher level of adaptive functioning. A positive change from baseline indicates an improvement in adaptive functioning. Composite V-scores have a mean (50th percentile) of 100 and a standard deviation (SD) of 15.
Time Frame: Baseline, Week 10
Population: ITT population: all randomized participants who received at least one dose of study drug and had at least one post-baseline assessment for at least one efficacy variable irrespective of compliance and protocol violations. Here "Overall number of participants analyzed, N" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil HCl | Placebo
Number analyzed (Participants) | 61 | 65
score on a scale
  Baseline | 83.1 (15.5) | 85.7 (15.8)
  Mean change from baseline at Week 10 | 4.74 (9.2) | 4.22 (8.5)

2. Secondary Outcome: Mean Change From Baseline in V-Scale Composite Score (Sum of 9 Sub-domains) of Vineland Adaptive Behavior Scales Second Edition-Parent Caregiver Rating Form (VABS-II/PCRF) at Week 4 and 10-Observed Cases (OC)
Description: The VABS-II/PCRF instrument was used in this study to assess 3 domains (each with 3 sub-domains): communication (sub-domains: receptive, expressive, writing), daily living skills (sub-domains: personal, domestic, community), and socialization (sub-domains: interpersonal relationships, play/leisure time, coping skills). Raw scores (2=always present, 1=sometimes present, 0=seldom or never present) rated by the parent/caregiver from each sub-domain were converted to standardized scores called V-scores, which are based on age and a national sample of normal children. Each sub-domain v-scale score ranged from 1 (weakness) to 24 (strength). V-scores for the 9 sub-domains were summed to obtain a composite V-score ranging from 9 to 216. Higher scores indicate a higher level of adaptive functioning. A positive change from baseline indicates an improvement in adaptive functioning. Composite V-scores have a mean (50th percentile) of 100 and a SD of 15.
Time Frame: Baseline, Week 4 and Week 10
Population: ITT population: all randomized participants who received at least one dose of study drug and had at least one post-baseline assessment for at least one efficacy variable irrespective of compliance and protocol violations. Here "Overall number of participants analyzed, N" signifies participants who were evaluable for this outcome measure. Here "Number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil HCl | Placebo
Number analyzed (Participants) | 61 | 65
score on a scale
  Baseline | 83.1 (15.5) | 85.7 (15.8)
  Mean change from baseline at Week 4: number analyzed (Participants) | 54 | 60
  Mean change from baseline at Week 4 | 1.5 (6.4) | 2.6 (8.5)
  Mean change from baseline at Week 10: number analyzed (Participants) | 55 | 63
  Mean change from baseline at Week 10 | 5.1 (9.6) | 4.2 (8.6)

3. Secondary Outcome: Mean Change From Baseline in Test of Verbal Expression and Reasoning (TOVER) Total Score at Week 4 and 10-OC
Description: The TOVER is a participant-performance-based measure of expressive language function and verbal reasoning in response to questions about a series of stylized pictures showing identifiable scenarios. The 64-item test was specifically designed to assess language function in children and adults with down syndrome (DS) across a broad range of functional ability. The test used 23 multi-colored pictures to stimulate verbal responses to questions. The test was short (completed in 15 minutes) and fast-paced (2 to 4 questions per picture). Total score ranging from 0 to 64, was derived from 64 questions, where higher score indicates better functional ability.
Time Frame: Baseline, Week 4 and Week 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil HCl | Placebo
Number analyzed (Participants) | 62 | 64
score on a scale
  Baseline | 20.7 (12.2) | 21.6 (11.4)
  Mean change from baseline at Week 4: number analyzed (Participants) | 56 | 59
  Mean change from baseline at Week 4 | 1.2 (6.4) | 0.9 (8.5)
  Mean change from baseline at Week 10: number analyzed (Participants) | 56 | 62
  Mean change from baseline at Week 10 | 2.6 (6.2) | 1.9 (5.5)

4. Secondary Outcome: Mean Change From Baseline in Test of Verbal Expression and Reasoning (TOVER) Total Score at Week 10-LOCF
Description: The TOVER is a participant-performance-based measure of expressive language function and verbal reasoning in response to questions about a series of stylized pictures showing identifiable scenarios. The 64-item test was specifically designed to assess language function in children and adults with DS across a broad range of functional ability. The test used 23 multi-colored pictures to stimulate verbal responses to questions. The test was short (completed in 15 minutes) and fast-paced (2 to 4 questions per picture). Total score ranging from 0 to 64, was derived from 64 questions, where higher score indicates better functional ability.
Time Frame: Baseline, Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil HCl | Placebo
Number analyzed (Participants) | 62 | 64
score on a scale
  Baseline | 20.7 (12.2) | 21.6 (11.4)
  Mean change from baseline at Week 10 | 2.4 (6.0) | 2.1 (5.5)

ADVERSE EVENTS:
Time Frame: Baseline up to 10 months
Arm/Group | Donepezil HCl | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/65
Other Adverse Events (participants affected / at risk) | 45/64 | 42/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil HCl (N=64) | Placebo (N=65)
Gastroenteritis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil HCl (N=64) | Placebo (N=65)
Abdominal pain, upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 11 | 10
Fecal incontinence (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 8 | 2
Fatigue (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 2
Bronchitis (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 1 | 3
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 4
Pharyngitis (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Viral infection (Infections and infestations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Headache (Nervous system disorders) | 5 | 2
Lethargy (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other